CLINICAL TRIAL: NCT05973448
Title: A Pragmatic Crossover Trial to Test the Effectiveness of a Novel Lighting System to Reduce Nighttime Falls in Persons With Alzheimer's Disease and Related Dementias
Brief Title: The Nightlight Falls Prevention Study
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: 22-1162; 1R01AG075010-01 (NIH)
Record Dates: First submitted 2023-07-21; First posted 2023-08-02 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Aging; Alzheimer Disease; Dementia Alzheimers; Dementia of Alzheimer Type; Fall Injury
Keywords: Aging; Alzheimer's Disease; Alzheimer's Disease Related Dementias; Assisted Living; Fall Injury
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Each participating community will have approximately 8-12 enrolled residents with ADRD. The AL communities will be randomized to four treatment sequences over the course of one year that define the order of the lighting intervention delivered across four 3-month (90 day) periods (N=335 residents). This design requires that the lights be turned on or off some periods, which will be done by research staff during scheduled visits. The four treatment sequences are chosen such that each resident receives control (C) lighting in two periods and novel lighting (L) in two periods and no more than 2 lighting changes. The four sequences are: CCLL, CLLC, LCCL, LLCC. There are no "washout" periods between the lighting conditions.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Lighting Sequence 1: CCLL (Other): In this arm, the participant will receive the control lighting condition (C) for the first two quarters (180 days) and then crossover to the novel lighting condition (L) for the last two quarters (180 days).
  Q1 - Control lighting Q2 - Control lighting Q3 - Novel lighting Q4 - Novel lighting
  Interventions: Other: Novel Lighting Condition; Other: Control Lighting Condition
- Lighting Sequence 2: CLLC (Other): In this arm, the participant will receive the control lighting condition (C) for the first quarter (90 days) and then crossover to the novel lighting condition (L) for the next two quarters (180 days) and finally crossover again to the control condition (C) for the last quarter (90 days).
  Q1 - Control lighting Q2 - Novel lighting Q3 - Novel lighting Q4 - Control lighting
  Interventions: Other: Novel Lighting Condition; Other: Control Lighting Condition
- Lighting Sequence 3: LCCL (Other): In this arm, the participant will receive the novel lighting condition (L) for the first quarter (90 days) and then crossover to the control lighting condition (C) for the next two quarters (180 days) and finally crossover again to the novel condition (L) for the last quarter (90 days).
  Q1 - Novel lighting Q2 - Control lighting Q3 - Control lighting Q4 - Novel lighting
  Interventions: Other: Novel Lighting Condition; Other: Control Lighting Condition
- Lighting Sequence 4: LLCC (Other): In this arm, the participant will receive the novel lighting condition (L) for the first two quarters (180 days) and then crossover to the control lighting condition (C) for the last two quarters (180 days).
  Q1 - Novel lighting Q2 - Novel lighting Q3 - Control lighting Q4 - Control lighting
  Interventions: Other: Novel Lighting Condition; Other: Control Lighting Condition

INTERVENTIONS:
Other: Novel Lighting Condition — Horizontal and vertical lights over a doorway visible from the bed
  Other Names: Indicated in sequence by "L"
Other: Control Lighting Condition — Standard night light plugged into wall socket
  Other Names: Indicated in sequence by "C"

SUMMARY:
This project will test the effectiveness of a novel intervention consisting of unobtrusive, low-intensity, horizontal and vertical lights that outline the bathroom or entry way doorframe in residents' rooms and provide visual cues to promote postural stability. Specifically, this pragmatic crossover trial will enroll 335 assisted living residents with dementia and follow them for one year, comparing the incidence of nighttime falls during the lighting condition to the incidence of falls during the control condition; secondarily, it will determine whether and to what extent the intervention effect is modified by resident- and environmental-level risk factors, and satisfaction with the lighting system.

DETAILED DESCRIPTION:
Falls are the primary cause of fatal and non-fatal injuries among persons 65 years of age and older. Dementia is a major risk factors for falls, and assisted living (AL) communities are the primary provider of residential care for ambulatory older adults with dementia, making AL a critical setting in which to reduce falls. Forty-two percent of the more than 811,000 AL residents across the U.S. have moderate or severe dementia, 84% are ambulatory, and more than a third experience a fall in a six-month period, putting them among the 15% of AL residents who suffer a hip fracture or other serious fall-related injury each year. Falls are responsible for one-third of all hospitalizations of AL residents, and the resulting injuries may lead to a cascade of events, including worsening function, nursing home transfer, and death.

A significant number of these falls occur in the bedroom during the evening and night, when AL staff are not present, thereby limiting their ability to intervene. However, the cause of many of these falls -- impaired nighttime vision and related postural instability -- suggests a promising avenue for intervention.

This project will test the effectiveness of a novel intervention consisting of unobtrusive, low-intensity, horizontal and vertical lights that outline the bathroom or entry way doorframe in residents' rooms and provide visual cues to promote postural stability. The lighting system is particularly attractive and pragmatic because it is low cost, requires no staff involvement, and can be easily installed in new buildings or retrofitted to existing buildings.

The study investigators recently completed a NIH R21 exploratory/developmental randomized crossover trial of this system and found a 34% decrease in falls due to a novel lighting intervention. This NIH R01 project will build on that preliminary effort; if the results are as promising as suggested, this pragmatic passive lighting system has the potential to reduce falls and related sequelae for countless persons with Alzheimer's disease and related dementias, and to become a new standard of care.

The intervention being tested is the effectiveness of a novel intervention consisting of unobtrusive, low-intensity, horizontal and vertical lights that outline the bathroom or entry way doorframe in assisted living (AL) residents' rooms in preventing night time falls. The trial will enroll 335 AL residents with Alzheimer's disease and related dementias (ADRD) from 36 assisted living communities. The lighting will be installed in the rooms of all 335 enrolled AL residents and compared to standard nightlights (control condition). Using a randomized crossover trial design, subjects will be examined under both conditions over one year. The trial will enroll 36 communities over the course of three years. Falls will be measured using SafelyYou, a fall detection system that uses video cameras and artificial intelligence to detect falls in resident rooms while maintaining resident privacy."

ELIGIBILITY:
Inclusion Criteria:

* Has a diagnosis of dementia
* Lives in a participating AL community
* Not blind
* Not on hospice and in a worsening state
* Not expected to die or transfer during the next 6 months
* Reside in a private room; or reside in a shared room if

  1. one resident is male and one is female and both are participating in the project, or
  2. they are of any gender, as long as there is a wall divider between their bedrooms
* Do not have an overnight sitter in the room every night

Exclusion Criteria:

• None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 335 (Estimated)
Dates: Start 2023-07-28 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Falls incidence density ratio | At study completion (one year)
  (Number of falls/Number of Nights Novel) / (Number of falls/Number of Nights Control)

CONTACTS AND LOCATIONS:
Overall Officials: Sheryl Zimmerman, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
With the exception of the falls video clips, all other individual participant data collected during the trial will be shared after deidentification.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication.
Access Criteria: An investigator who proposes to use the data must have approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and execute a data use/sharing agreement with UNC.